

## Informed consent form

# Digital Detox Study

A randomized controlled trial with two unblinded, parallel arms assessing the effect of reducing smartphone screen time on mental health

Authors: Katja Haider, BA MSc,

Prof. Dr. Christoph Pieh

Version: 02

Clinical trial phase: n.a.

Release date: March 25, 2025



#### **Digital Detox Study**

#### 1) Information about the study

The Digital Detox study is conducted at the University for Continuing Education Krems, Department for Psychosomatic Medicine and Psychotherapy, and is led by Prof. Dr. Christoph Pieh.

The aim of the study is to investigate the effects of reducing smartphone screen time on mental health. For this purpose, there is an intervention group and a control group, to which you will be randomly assigned after completing the first questionnaire. The intervention group will start with a three-week intervention phase in which smartphone screen time should not exceed two hours per day. The control group continues to use their smartphone as usual during this time. After the three-week intervention, the intervention group also uses their smartphone again without restriction.

Mental health questionnaires are provided to both groups before and after the intervention and at a follow-up point (3 weeks after the end of the intervention), as well as a short questionnaire twice during the intervention. You will, of course, receive further instructions from the study team on time regarding what is to be done at the respective points in time.

The data on mental health and screen time are collected in the ESMira app (Karl Landsteiner University of Health Sciences, Dr.-Karl-Dorrek-Str. 30, 3500 Krems). The questionnaires collect information about your age, gender, highest level of education, educational/professional status, place of residence, mental health, exercise, and smartphone use. Your data will be collected and processed pseudonymously. It is not possible to draw conclusions about you, even when combining several characteristics. Study results will only be published in aggregated form.

Anonymous contact with the study team with questions and concerns about the study is possible via the chat function in the ESMira app. In addition, the study team can be reached by email at <a href="mailto:istokay@donau-uni.ac.at">istokay@donau-uni.ac.at</a>.

Your participation in the study is voluntary. You can revoke your consent at any time without giving reasons and discontinue the study. All study staff are subject to professional confidentiality and are bound to data secrecy.

### 2) Data protection declaration

Responsible in accordance with Article 4(7) of the DSGVO: University for Continuing Education Krems, Department for Psychosomatic Medicine and Psychotherapy, Contact person: Prof. Dr. Christoph Pieh, Dr.-Karl-Dorrek-Straße 30, 3500 Krems an der Donau, +43 2732 893-2530 or christoph.pieh@donau-uni.ac.at

Data protection officers: Dr. Daniel Stanonik LL.M., attorney, and KINAST Rechtsanwaltsgesellschaft mbH, represented by Dr. Karsten Kinast LL.M., attorney, in mutual representation datenschutz@donau-uni.ac.at or +43 2732 8930



Legal basis: Art. 85, 89 in conjunction with Art. 6 (1) lit a DSGVO in conjunction with § 3 Z 1, 7 & 8 Universitätsgesetz (UG)

The recipients of the raw research data are the scientific staff of the Center for Mental Health Research at the University for Continuing Education Krems.

Storage period: The pseudonymized raw research data will be stored until the end of the study period.

Legal information: To make use of your rights to information, deletion, etc. in accordance with Art. 15 - 20 DSGVO, please contact the above-mentioned contact person or, subsidiarily, the data protection officer. Due to a lack of identifiability, your rights may be restricted without the provision of further information in accordance with Art. 11 DSGVO.

Please direct any complaints to the Austrian data protection authority: www.dsb.gv.at

| I have read the information about the study and the data protection declaration and agree to par- |
|---|
| ticipate in the study and to the processing of my personal data in this context. This consent can |
| be revoked at any time in the future. |